CLINICAL TRIAL: NCT03384355
Title: Ecchymosis and Coldness in Patients With Varicose Vein: Multicenter Study of Modified VEIN-Sym QoL Assessment
Brief Title: Ecchymosis and Coldness in Patients With Varicose Vein
Acronym: VEIN-COLD
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Vascular and Molecular Cardiology Society (Other)
Responsible Party: Sponsor
Other Study IDs: Vasmol003
Record Dates: First submitted 2017-12-18; First posted 2017-12-27 (Actual); Last update posted 2017-12-27 (Actual); Status verified 2017-12

CONDITIONS: Varicose Veins; Chronic Venous Insufficiency; Symptoms and General Pathology
Keywords: varicose veins; chronic venous disease; ecchymosis; symptoms
MeSH Terms: conditions — Varicose Veins; Pathological Conditions, Signs and Symptoms; Ecchymosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (7):
- Class 0: no visible or palpable varicose veins
- Class 1: telengiectasia ( thread veins, spider veins, broken veins)
- Class 2: varicose veins
- Class 3: edema
- Class 4: skin changes (pigmentation, eczema, lipodermatosclerosis, atrophie blanche)
- Class 5: healed venous ulcer
- Class 6: active venous ulcer

SUMMARY:
In this prospective, observational study, the investigators aim to investigate the symptoms of varicose vein patients.

DETAILED DESCRIPTION:
Chronic venous disease is very common in all over the world and affects both the mortality and morbidity depending on the effected vascular territory. It is often overlooked by healthcare professionals due to the underestimation of the prevalence and impact of the disease. It represents a spectrum of conditions varying from simple telangiectasia or reticular veins to skin fibrosis and venous ulceration. The main clinical characteristics are dilated veins, edema, leg pain, and cutaneous alterations in the legs. Varicose veins are dilating superficial veins, which become more tortuous and enlarged, continuously.

Chronic venous disease affects the life quality of patients suffering from the disease, which can be measured with quality-of-life reports. Venous Insufficiency Epidemiological and Economic Study-Quality of Life/Symptoms (VEINES-QoL/Sym) questionnaire is a patient based, designed for self-completion instrument to measure both the symptom severity and quality of life. VEINES-QOL measures life quality and VEINES-Sym provides an overall estimate of CVD symptom frequency. From the practitioners daily knowledge of patients with varicose veins, there is a significant proportion of varicose vein patients also suffering from symptoms such as coldness and ecchymosis. In this context, the investigators aim to investigate the symptoms of participants with varicose vein using the VEINES-Sym questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* acceptance of inclusion
* aged between 18-75 years

Exclusion Criteria:

* < 18 year old
* > 75 year old
* malignancy
* active infection
* hematological disease (severe anemia, leukemia, polistemia vera, sickle cell disease)
* collagen tissue disease
* severe decompensated heart failure (ejection fraction < 40%)
* cor pulmonale
* rheumatoid arthritis
* degenerative arthritis
* history of lower extremity orthopedic surgery
* lombar disk hernia
* history of coronary artery by-pass surgery
* severe psychiatric and neurological disease (parkinson disease, schizophrenia, bipolar disease, alzheimer disease, etc.)
* peripheral arterial disease ( history of interventional procedure, claudication, active ischemic complaints)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients admitting to cardiology and/or cardiovascular surgery outpatient clinics and do not match the exclusion criteria
Sampling Method: Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2018-01 (Estimated); Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Venous Insufficiency Epidemiological and Economic Study- Symptom score evaluation | baseline
  Venous Insufficiency Epidemiological and Economic Study-Quality of Life/Symptoms (VEINES-QoL/Sym) questionnaire is a patient based, designed for self-completion instrument to measure both the symptom severity and quality of life. VEINES-QOL measures life quality and VEINES-Sym provides an overall estimate of CVD symptom frequency. Lower VEINES-Sym scores indicate more severe symptoms and higher VEINES-QoL/Sym scores indicate better QoL.VEINES-Sym consists of ten items including nine venous symptoms (heavy legs, aching legs, swelling, night cramps, heat/burning sensation, restless legs, throbbing, itching and tingling sensation) in five different frequencies (1=everyday, 2= several times a week, 3= about once a week, 4= less than once a week, 5= never) and leg pain rated on a six-point scale of intensity (1 = very severe, 2= severe, 3 =moderate, 4 = mild, 5 =very mild, 6= none).

SECONDARY OUTCOMES:
Evaluation of additional symptoms | baseline
  Evaluation of additional symptoms (coldness and ecchymosis)
CEAP (clinical, etiological, anatomical and pathological) clinical classification | baseline
  CEAP clinical classification is an physical examination based scale to measure the severity of chronic venous disease: grade 0, no visible signs of venous disease; grade 1, telangiectasias or reticular veins; grade 2, varicose veins; grade 3, edema; grade 4, skin changes due to CVD; grade 5, skin changes with healed ulceration; and grade 6, skin changes with active ulceration.

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet Ileri, MD, Study Chair — Ankara City Hospital Bilkent

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Ozturk S, Yetkin E. Identifying symptoms in chronic venous diseases. Eur J Obstet Gynecol Reprod Biol. 2016 Aug;203:331. doi: 10.1016/j.ejogrb.2016.04.011. Epub 2016 Jun 23. No abstract available. PMID 27401694
- [Result] Yetkin E, Ileri M. Dilating venous disease: Pathophysiology and a systematic aspect to different vascular territories. Med Hypotheses. 2016 Jun;91:73-76. doi: 10.1016/j.mehy.2016.04.016. Epub 2016 Apr 11. PMID 27142148
- [Result] Yetkin E. Hemorrhoid, internal iliac vein reflux and peripheral varicose vein: Affecting each other or affected vessels? Phlebology. 2015 Mar;30(2):145. doi: 10.1177/0268355514565196. Epub 2014 Dec 19. No abstract available. PMID 25527517
- [Result] Yetkin E, Öztürk S and Ileri M. Varicose Vein And Ecchymosis: A Case Report. International Archives of Medicine. 2017; 10.
- [Result] Yetkin E. Complexity of venous symptoms. Phlebology. 2016 Mar;31(2):147. doi: 10.1177/0268355515574152. Epub 2015 Feb 19. No abstract available. PMID 25700552
- [Result] Yetkin E. Images in Vascular Medicine. A new or overlooked finding of varicose veins: Ecchymosis. Vasc Med. 2016 Feb;21(1):75-6. doi: 10.1177/1358863X15607654. Epub 2015 Oct 5. No abstract available. PMID 26443802
- [Result] Yetkin E, Ileri M, Waltenberger J. Ecchymosis: A novel sign in patients with varicose veins. Clin Hemorheol Microcirc. 2018;68(4):413-419. doi: 10.3233/CH-170320. PMID 29660929